CLINICAL TRIAL: NCT06854562
Title: The Effectiveness of Using a Therapeutic Robot to Alleviate Hospitalization Stress Among Children in Intensive Care Units: A Randomized Controlled Trial
Brief Title: Therapeutic Robots for Alleviating ICU Stress in Children
Acronym: NYMCTU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-02-017C
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Intensive Care Units
Keywords: Therapeutic Robot; Pediatric Intensive Care Unit (PICU); School-age Children; Adolescents; Hospitalization Stress Response
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Robot Seal Therapy (Experimental): Arm 1 (Robot Seal Therapy):
  Description: Children in this group will interact with a therapeutic robot seal designed to alleviate stress and provide emotional comfort. The robot seal will be used as a companion during their stay in the Pediatric Intensive Care Unit (PICU) to reduce feelings of anxiety and stress.
  Interventions: Behavioral: Therapeutic Robot Intervention
- Arm 2: Toy Seal Therapy (Experimental): Arm 2 (Toy Seal Therapy):
  Description: Children in this group will engage with a toy seal as a comforting object. The toy seal will be used to help children cope with the hospital environment and reduce stress during their PICU stay.
  Interventions: Behavioral: Toy Seal Intervention
- Arm 3: Standard Care (Active Comparator): Arm 3 (Standard Care):
  Description: Children in this group will receive standard care and routine interventions provided by healthcare professionals in the PICU without the use of additional therapeutic devices.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Therapeutic Robot Intervention — This intervention involves the use of a therapeutic robot seal, PARO, to interact with pediatric patients in the Pediatric Intensive Care Unit (PICU). The intervention is designed to alleviate stress and anxiety in children during their hospital stay. The robot provides emotional support by engaging in 30-minute sessions, where children can interact with the robot, give it a name, and express their emotions. The therapeutic interaction is repeated twice on consecutive days.
  Other Names: Robot Seal Therapy
  Arms: Arm 1: Robot Seal Therapy
Behavioral: Toy Seal Intervention — In this group, children interact with a plush toy seal. The plush seal is used to provide emotional comfort and reduce anxiety during their stay in the PICU. The interaction happens over two consecutive days for 30 minutes per session.
  Arms: Arm 2: Toy Seal Therapy
Behavioral: Standard Care — Children in this group will receive standard care and routine interventions provided by healthcare professionals in the PICU, without the use of therapeutic robots or plush toys.
  Arms: Arm 3: Standard Care

SUMMARY:
The purpose of this study is: (a) to examine the changes in anxiety, depression symptoms, and positive/negative emotions before and after the intervention, as well as before discharge from the intensive care unit (ICU) in the experimental group (using the therapeutic robot PARO), the control group (using a stuffed seal), and the comparison group (receiving standard care). (b) To compare the effectiveness in relieving anxiety, depression symptoms, and positive/negative emotions among the experimental group, control group, and comparison group for ICU pediatric and adolescent patients in the school-age period.

The research questions addressed in this study are:

1. What are the changes in anxiety, depression symptoms, and negative emotions before and after the intervention in the experimental group?
2. What are the changes in anxiety, depression symptoms, and negative emotions before and after the intervention in the control group?
3. What are the changes in anxiety, depression symptoms, and negative emotions before and after the intervention in the comparison group?
4. What is the effectiveness in reducing anxiety after the intervention among the experimental group, control group, and comparison group?
5. What is the effectiveness in alleviating depression symptoms after the intervention among the experimental group, control group, and comparison group?
6. What is the effectiveness in reducing negative emotions and increasing positive emotions after the intervention among the experimental group, control group, and comparison group?

DETAILED DESCRIPTION:
Children and adolescents in the intensive care unit (ICU) often find themselves in a confined, lonely environment due to changes in their health status. Their cognitive and self-concept development is not yet mature, making them prone to developing defense mechanisms and suppressing emotions. This can lead to noncompliance with treatment in an attempt to regain a sense of control, which further triggers negative emotions and affects their condition. Therapeutic robots, through human-robot interaction and a cute appearance, help alleviate stress and improve positive emotions by providing companionship and interaction. However, there is currently a lack of research on the effectiveness of therapeutic robots in ICU settings for hospitalized children and adolescents, which motivates this study. This research aims to explore the effectiveness of using therapeutic robots to alleviate the hospitalization stress of school-age children and adolescent patients in the ICU. The study will be conducted at the pediatric ICU of a medical center in northern Taiwan, and participants will include 8 to 18-year-old school-age children and adolescents who are hospitalized in the ICU. Participants will be randomly assigned into the experimental group, control group, and comparison group. The experimental group will use the therapeutic robot PARO as an intervention strategy, the control group will use a stuffed seal, and the comparison group will receive standard care. During the study, the Multidimensional Anxiety Scale for Children, the Children's Depression Inventory, and the Positive and Negative Emotion Scale will be used to measure the stress response of the three groups before the intervention, after the intervention, and before discharge from the ICU. Semi-structured interviews will be conducted using the triangulation method. Quantitative data will be analyzed using covariance analysis and generalized estimating equations, while qualitative data will be analyzed using content analysis. This study aims to develop an intervention measure to alleviate hospitalization stress in children in the ICU and evaluate its effectiveness. It is expected that through the interactive communication concept of the therapeutic robot, the social abilities of school-age children and adolescents will be enhanced, leading to an improvement in their positive emotional expression and promoting their psychological health.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the intensive care unit (ICU).
2. Age range for enrollment is 8 to 18 years.
3. Able to stay awake and respond.
4. Able to communicate in Mandarin or Taiwanese.
5. Have been informed and have agreed to participate in the study.

Exclusion Criteria:

1. Patients with a pacemaker.
2. Patients who require isolation according to hospital infection control regulations.
3. Patients with wounds that continue to ooze under the gauze covering.
4. Patients experiencing vomiting symptoms within the past 24 hours.
5. Patients assessed by a physician to be in a life-threatening condition.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Before the intervention, immediately after the intervention, and before discharge from the intensive care unit (ICU).
  The Multidimensional Anxiety Scale for Children will be used to measure the patient's anxiety. This scale includes multiple dimensions, typically assessing emotional, behavioral, and physiological responses. Each dimension consists of several questionnaire items, rated on a Likert scale with a range from 0 to 3, and includes a total of 39 items. The total score correlates with the level of anxiety, with higher scores indicating higher anxiety. This scale provides a comprehensive assessment of the child's anxiety from multiple perspectives.
Depression | Before the intervention, immediately after the intervention, and before discharge from the intensive care unit (ICU).
  The Children's Depression Inventory (CDI) - Short Version is a screening tool used to assess the level of depression in children and adolescents. It consists of a shortened set of items that evaluate emotional, behavioral, and cognitive symptoms related to depression. The scale typically includes 12 items, each rated on a Likert scale, with higher scores indicating more severe symptoms of depression. The tool provides a quick yet effective measure of depressive symptoms in children, helping to identify those who may need further evaluation or intervention.
Positive and Negative Affect | Before the intervention, immediately after the intervention, and before discharge from the intensive care unit (ICU).
  The Positive and Negative Affect Schedule (PANAS) is a psychological tool used to measure both positive and negative emotional states in individuals. It consists of two subscales: one assessing positive affect (PA) and the other assessing negative affect (NA). Each subscale includes a list of emotional terms, with participants rating the extent to which they have experienced these emotions during a specified time frame (e.g., the past week, day, or moment). The items are rated on a Likert scale, usually ranging from 1 (very slightly or not at all) to 5 (extremely). Higher scores on the positive affect subscale indicate a higher level of positive emotions, while higher scores on the negative affect subscale indicate a higher level of negative emotions. PANAS is commonly used in both research and clinical settings to assess mood, emotional well-being, and emotional responses to various stimuli or interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Yi Ke, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: No